CLINICAL TRIAL: NCT02975232
Title: Supermarket Science: Multipronged Approaches to Increasing Fresh, Frozen and Canned Fruit and Vegetable Purchases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Michele Polacsek, Associate Professor, University of New England
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-68001-24961
Record Dates: First submitted 2016-11-16; First posted 2016-11-29 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Obesity
Keywords: nutrition disparities; SNAP population; behavioral economics; retail setting; point of purchase education; pediatric obesity; rural population; fruit and vegetable purchases; fruit and vegetable consumption
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): F&V economic incentive with Cooking Matters store tour
  Interventions: Behavioral: F&V economic incentive; Behavioral: Cooking Matters Store Tour
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: F&V economic incentive — 50% off eligible fresh, frozen and canned fruits and vegetables (up to $10/day)
  Arms: Treatment
Behavioral: Cooking Matters Store Tour — Participants will be asked to attend one Coking Matters store tour during January or February 2017
  Arms: Treatment

SUMMARY:
Through research, education and extension, this project will promote fruit and vegetable (F&V) purchases and consumption by families in under-resourced communities, thus reducing health disparities, improving human nutrition, and preventing unhealthy weight gain among children. Specifically, this project aims to evaluate the success of promoting F&V purchases among low- income and Supplemental Nutrition Assistance Program (SNAP)-eligible families and children living in a rural Maine community through a double value coupon, supermarket- based incentive program combined with Cooking Matters at the Store education. Education and extension efforts based on the study findings will contribute to meeting USDA Childhood Obesity Prevention Challenge Area Goals of generating new knowledge; developing, assessing and expanding effective interventions; and increasing the number of skilled and informed professionals and consumers to address the complex problem of childhood obesity. The research team will partner with a large national retail grocery chain (Hannaford Brothers), Cooking Matters, University of Maine Cooperative Extension, eXtension Communities of Practice, Maine SNAP-Ed, and The Food Trust to accomplish the project objectives.

DETAILED DESCRIPTION:
Through research, education and extension, this project will promote fruit and vegetable (F&V) purchases and consumption by families in under-resourced communities, thus reducing health disparities, improving human nutrition, and preventing unhealthy weight gain among children. Specifically, this project aims to evaluate the success of promoting F&V purchases among low- income and SNAP-eligible families and children living in a rural Maine community. The project will use a multipronged approach in the supermarket setting, including implementation methods from the highly effective, double value coupon incentive program used at farmers' markets, as well as the Cooking Matters at the Store educational program to incentivize the purchase and consumption of fresh produce, and healthful frozen and canned F&V (without syrup or salt), nutrient-rich and affordable year- round alternatives to fresh produce.

Education and extension efforts based on the study findings will contribute to meeting United States Department of Agriculture (USDA) Childhood Obesity Prevention Challenge Area Goals of generating new knowledge; developing, assessing and expanding effective interventions; and increasing the number of skilled and informed professionals and consumers to address the complex problem of childhood obesity. The project team will partner with a large national retail grocery chain (Hannaford Brothers), Cooking Matters, University of Maine (UMaine) Cooperative Extension, eXtension Communities of Practice, Maine SNAP-Education (SNAP-Ed), and The Food Trust to accomplish its objectives.

Methods:

Research Strategy: The study will enroll 600 shoppers (and assume 70% retention, with an initial N of 600: n=210 per study arm) entering the store in months 6-7. If a customer has interest in participating and meets enrollment criteria (having a child between ages 2 and 18 years of age living in the household, and use of the Hannaford store as the primary grocery shopping venue), then the customer will be asked to enroll. At enrollment, research assistants will obtain informed consent, instruct participants about how to join "MyHannaford" in order to receive a unique study ID for tracking of all purchases, and give participants a MyHannaford "study loyalty" card and Guiding Stars information. A short survey will be administered to collect information about demographics (age, gender, family size, ethnicity), shopping habits (e.g. percent of total grocery shopping done at this Hannaford and person doing most of the shopping in the household), best method to communicate incentive changes once randomization has occurred, and F&V promotion reminders (e.g. text, email, mail), SNAP eligibility, and SNAP participation. Through the loyalty card and study ID, all participants will receive a 5% discount on all purchases at the participating Hannaford store during months 6-16 of the project.

Semi-quantitative Food Frequency Questionnaire (FFQ): The FFQ consists of approximately 130 food items and is regularly updated to account for changes in the availability of foods. At baseline and post intervention, participants will be emailed a link to the FFQ administered online through Qualtrics, which will take approximately 20 minutes to complete. Participant who complete the survey will be emailed an e-gift card. Participants will be asked to identify one index child in the household closest to the age range of 6-10 yrs (where children may be most receptive and influenced by parents eating patterns). Participants will be provided an excerpted section of the FFQ with only F&V listed for the respondent to complete, representing the child's average at-home consumption.

Randomization: After the 2-month baseline run-in period, study participants will be randomly assigned to double value coupon incentive program + Cooking Matters intervention, or control.

Intervention arm: Participants randomized to the intervention arm will receive 2 for 1 F&V (double value max $10 benefit per household per shopping day) for purchasing either fresh or 2 and 3-star-rated frozen and canned F&V in months 10-13. These will be confirmed by linking UPC codes with qualifying foods. All discounts (5% and incentive) will be given at checkout through the use of the loyalty card with assigned study ID. Participants will be asked to register and attend at least 1 of 5 Cooking Matters at the Store education program tours scheduled during the first two months of the intervention period (months 10-11). On the day and time of the Cooking Matters at the Store tour, there will be a Cooking Matters table set up in the entrance of the lobby. All shoppers at the store, regardless of study participation, are invited to join the tour. Study participants will be asked to sign in with their name or study ID (for tracking purposes) and pick up their "passport" (a card that must be stamped at each station in order to complete the tour) at the table in the lobby. The passport must have stamps from each station in order for the participant to receive a Hannaford gift card and participate in the $10 challenge (buying a healthy meal for a family of four for under $10).

Control arm: Participants assigned to the control arm will not be eligible for F&V incentives and will not be asked to attend Cooking Matters at the Store.

Post-intervention, all participants will continue to receive the 5% discount and we will continue tracking purchases for three additional months (months 14-16) using the study ID to examine retention of purchasing habits. During month 14 (1 year after baseline assessment), participants will be emailed a link to the FFQ, including the child portion, to assess average daily intake over the previous year. Reminders to complete and return the FFQ will be sent by text.

Data and analysis plan--F&V Sales: Primary study outcomes will be compared within individuals (pre- to post-intervention), and between individuals (intervention and control arms). Cooking Matters education program attendance between intervention and control arms will be compared. Mixed effects generalized linear models will be used to control for sex, primary household shopper, family size, month of purchase, and SNAP status (ineligible, eligible, enrolled).

Education and Extension Activities (post research):

Maine SNAP-Ed: The Maine SNAP-Ed program will contribute to education and extension efforts in years 3 and 4 of the grant by assisting with the development of resources, such as fact sheets and webinar trainings. Direct education classes will be used to disseminate resource materials developed through the grant. Maine SNAP-Ed can also help disseminate innovative approaches to work with supermarkets and grocers through their work with the USDA Food and Nutrition Service and the Association of SNAP Nutrition Education Administrators (ASNNA).

University of Maine Cooperative Extension: In year 3, UMaine Cooperative Extension staff will work to develop and finalize educational materials that will be used in project dissemination activities in year 4 of the project. In year 4, UMaine Cooperative Extension staff will provide two webinars for two different Maine audiences. One webinar will be conducted for Cooperative Extension's 4H Youth Development and nutrition staff, and the second will be delivered to Healthy Maine Partnership/SNAP-Ed staff. UMaine Extension Staff will also assist in creating and delivering an online training to both the eXtension Families, Food and Fitness, and Community Nutrition Education Communities of Practice. Additionally, project outcomes will be presented at the national Expanded Food and Nutrition Education Program annual meeting in Washington, DC. The Community Nutrition Education Program Community of Practice has also agreed to serve as host for materials developed through this project.

The Food Trust: In year 3, The Food Trust will prepare for education and extension efforts in year 4. The Food Trust will use its experience as a national partner on a variety of healthy food access policy and program efforts at the national, state, and local levels. In year 4, The Food Trust will work with UNE and partners to lead the development of an educational toolkit targeted at academic institutions, professional associations, and industry partners (e.g. retail chains and industry associations) to support development and enhancement of curricula and corresponding materials related to promoting healthy shopping behaviors in low-income populations.

University of New England (UNE): The University of New England is in the late planning stages of a Bachelor of Science in Nutrition degree. The study will provide a unique opportunity for undergraduate students to be involved in the community on issues related to food access among low-income populations.

Target Audiences Target audience for the research component: English-speaking, rural Maine families with at least one child under 18 years of age living in the household, regularly shopping at the study Hannaford store location. Westbrook is a low-income (median household income was $44,465 compared to the state level of $48,453 in 2013), mostly white (92% white in 2013), rural community in Southern Maine. The study Hannaford store in Westbrook has a high SNAP-user customer base ($90+Million in sales and 10% SNAP sales representing ~20% of UPC eligible sales in 2014).

Target audience for education and extension components: The Maine SNAP-Ed program staff; Maine Cooperative Extension staff and partners, The Nutrition Education Program Community of Practice, Food Trust staff and partners, University of New England Nutrition Program staff and faculty and low income families shopping in supermarket settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* at least one child in household aged 18 or younger
* at least 50% of grocery shopping done at study store location
* active cell phone accepting text messages
* active email address

Exclusion Criteria:

* non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2016-04; Primary Completion 2018-09 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Before discount spending (in dollars) on eligible fresh, frozen and canned F&V | through study completion, one year
  average change from baseline weekly and per transaction before discount spending (in dollars) on eligible fresh, frozen and canned F&V
nutrition behavior: shopper and 1 index child | at 1 month and up to 15 months
  change from baseline

OTHER OUTCOMES:
Frequencies of shopper nutrition behaviors practiced over the past week related to shopping and food preparation | at 1 month and up to 15 months
  self-reported nutrition behavior

CONTACTS AND LOCATIONS:
Overall Officials: Michele Polacsek, PhD MHS, Principal Investigator — University of New England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moran A, Thorndike A, Franckle R, Boulos R, Doran H, Fulay A, Greene J, Blue D, Block JP, Rimm EB, Polacsek M. Financial Incentives Increase Purchases Of Fruit And Vegetables Among Lower-Income Households With Children. Health Aff (Millwood). 2019 Sep;38(9):1557-1566. doi: 10.1377/hlthaff.2018.05420. PMID 31479362